CLINICAL TRIAL: NCT01313078
Title: Phase II Study of Clinical Activity of Pegaspargase in Women With Relapsed or Refractory Epithelial Ovarian Cancer, Fallopian Tube Cancer, and/or Primary Peritoneal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Elise C. Kohn, M.D./National Cancer Institute, National Institutes of Health
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 100028; 10-C-0028
Record Dates: First submitted 2011-03-09; First posted 2011-03-11 (Estimated); Results first posted 2012-09-12 (Estimated); Last update posted 2015-10-09 (Estimated); Status verified 2012-08

CONDITIONS: Ovarian Neoplasms; Fallopian Tube Neoplasms; Primary Peritoneal Neoplasms
Keywords: Ovarian Cancer; Fallopian Tube Cancer; Primary Peritoneal Cancer; Relapsed or Refractory; Pegaspargase; Pegylated L-Asparaginase
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms; Recurrence | interventions — pegaspargase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pegaspargase in women with cancer (Experimental): Pegaspargase 2000 IU/m^2 intramuscular or intravenously every 2 weeks
  Interventions: Drug: Pegylated L-Asparaginase

INTERVENTIONS:
Drug: Pegylated L-Asparaginase — Pegaspargase 2000 IU/m^2 intramuscular or intravenously every 2 weeks
  Other Names: Oncaspar

SUMMARY:
Background:

- The best treatment for ovarian and related female reproductive tract cancers is not yet known for patients whose disease has not responded to or has recurred after standard treatment. The cancer treatment drug pegaspargase (ONCASPAR (Trademark)), which works differently from standard chemotherapy, has been approved to treat leukemia and has been given to a small number of patient with ovarian and other types of cancer. Because pegaspargase may reduce the development of cancer cells and blood vessel cells that contribute to cancer growth and ability to spread, treatment with pegaspargase could shrink ovarian cancer tumors and help ovarian cancer patients live longer and with fewer symptoms from their disease.

Objectives:

- To evaluate the safety and effectiveness of pegaspargase in patients with recurrent or refractory ovarian cancer, fallopian tube cancer, and/or primary peritoneal cancer.

Eligibility:

- Women at least 18 years of age who have been diagnosed with epithelial ovarian cancer, fallopian tube cancer, or primary peritoneal cancer that has not responded to at least one operation, chemotherapy, and/or radiotherapy.

Design:

* Before the start of the study, participants will be screened with a medical history, blood tests, imaging scans of the affected areas, tumor biopsies, and other tests as directed by the study doctors.
* Participants will receive an infusion of pegaspargase on Day 1 and Day 15 of each 28-day cycle.
* Participants will have dynamic contrast-enhanced magnetic resonance imaging (DCE-MRI) at the start of the study, before beginning pegaspargase, and again 6 weeks into the treatment. This test will determine if pegaspargase is affecting blood flow to the cancer site.
* Participants will have a computed tomography scan or other imaging every other cycle (approximately every 8 weeks) to determine whether the therapy is affecting the cancer site.
* The treatment will be repeated as long as the participant tolerates the medication and his or her cancer is either steady or improving.

DETAILED DESCRIPTION:
Background:

* The bacterial enzyme L-asparaginase (L-ASP) catalyzes hydrolysis of asparagine to aspartate and is used to treat acute lymphoblastic leukemia (ALL).Studies demonstrated in vitro cytotoxic activity against solid tumor types including ovarian cancer.
* Our laboratory demonstrated L-ASP inhibits vascular remodeling and modulates heterotypic adhesion interactions between ovarian cancer cells and endothelial cells. Results indicate L-ASP has the ability to modify the local tumor microenvironment.
* Epithelial ovarian cancer requires neovascularization for growth and metastasis. Anti-angiogenesis agents show promise in treatment of recurrent disease.
* The pegylated form of L-ASP, pegaspargase, (Sigma Tau ONCASPAR (Trademark)) is shown to deplete serum levels of asparagine and is approved for ALL. ONCASPAR is in clinical trial with gemcitabine for pancreatic cancer and other solid tumors.
* Recommended dose of pegaspargase in ALL is 2,500 IU/m^2 every two weeks intramuscular (IM)/intravenous (IV). IM dosing of 2,000 IU/m^2 every two weeks has been studied in a phase I protocol with various solid tumors.
* Demonstration of safety and anti-angiogenic activity will lead to combination studies.

Primary Objectives:

* To preliminarily evaluate the anti-tumor activity of pegaspargase, 2,000 IU/ m^2 every two weeks intravenous (IV) (or intramuscular (IM)) and explore associations with toxicity and clinical outcome.
* To evaluate the safety of pegaspargase in patients with recurrent or refractory ovarian, fallopian tube, and/or primary peritoneal cancer.

Secondary Objectives:

* To explore changes in circulating angiogenic cytokines after treatment with pegaspargase.
* To measure apoptosis and proliferation in tumor (or malignant effusion) by protein array before and during therapy.
* To evaluate changes in tumor vascularity using dynamic contrast enhanced (DCE) magnetic resonance imaging (MRI).

Eligibility:

* Women with epithelial ovarian cancer, fallopian tube cancer, and/or primary peritoneal cancer that is persistent, relapsed and/or refractory to prior therapy.
* There is no limit to number of prior treatment regimens. Patients may not have previously received L-ASP.
* Women must have disease amenable to biopsy or malignant effusions (pleural effusion or ascites) that may be serially tapped.
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1, 2.
* Evidence of adequate end organ function and normal coagulation parameters (prothrombin time (PT), activated partial thromboplastin time (aPTT)).

Design:

* Women will receive 2,000 IU/m^2 of pegaspargase intravenously every two weeks in 28-day cycles until disease progression, excessive toxicity, or withdrawal from study.
* Biopsy of tumor and dynamic contrast-enhanced-magnetic resonance imaging (MRI) will be performed prior to starting pegaspargase (mandatory) and after 6 weeks of treatment (optional).
* Clinical outcome will be measured and correlated with biological endpoints.
* Research blood samples will be taken to assess changes in serum vascular endothelial growth factor (VEGF), interleukin-6 (IL6), and interleukin-8 (IL8).
* Blood will be collected to evaluate circulating endothelial cells.
* Patients will be seen in clinic every 4 weeks and outcome measured every other cycle.

ELIGIBILITY:
* INCLUSION CRITERIA:
* All patients 18 years and older with epithelial ovarian, fallopian tube, or primary peritoneal cancer that is persistent, relapsed or refractory to prior standard platinum and taxane-based therapy will be eligible. Tumor histology must be reviewed and confirmed by the National Cancer Institute (NCI) Laboratory of Pathology. Recurrent ovarian cancer is not a curable tumor. Patients who are platinum-sensitive and who, upon detailed informed consent, wish to consider this experimental regimen, will be considered.
* All patients must have measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) criteria. A sentinel lesion adequate for core biopsy through percutaneous route is ideal but not mandatory. Patients with a malignant pleural effusion or malignant ascites will be allowed to undergo a paracentesis or thoracentesis rather than core needle biopsy if the procedure may be performed safely.
* Patients must have a performance status of Eastern Cooperative Oncology Group (ECOG) = 0, 1, 2
* Patients must have adequate end organ function:

  * Absolute neutrophil count (ANC) greater than or equal to 1500/ mm^3
  * Platelets greater than or equal to 100,000/ mm^3
  * Serum creatinine less than or equal to 1.5 mg/dL, or if low, creatinine clearance greater than or equal to 60 mL/min
  * Total bilirubin less than or equal to 1.5 times the ULN (upper limit of normal) unless a history of Gilbert's disease.
  * Lipase and amylase less than or equal to 1.5 times the ULN
  * Transaminases (aspartate aminotransferase (AST), alanine aminotransferase (ALT)) less than or equal to 2.5 times the ULN
  * Fibrinogen greater than or equal to 0.75 times the LLN
  * Prothrombin time (PT), partial thromboplastin time (PTT), and International Normalized Ratio (INR) less than or equal to 1.5 times the ULN. Coagulation parameters must be drawn peripherally.
* Patients must be at least 4 weeks from previous therapy (chemotherapy, hormonal therapy, and radiation therapy, alternative therapy, investigational agents, or a major surgical procedure). Patients must be 6 weeks from carboplatin- or mitomycin C-containing therapy. Exceptions: Raloxifene will be allowed for bone health and bisphosphonate therapy will be allowed for the rare situation of bone metastasis.
* There is no limit to the number of prior regimens patients may have received for the treatment of ovarian cancer.
* Patients must have recovered from any toxicity related to prior cancer therapy to Common Terminology Criteria for Adverse Events (CTCAE) grade 1, except for stable peripheral neuropathy, which must have recovered to grade 2 or better, and grade 2 total white blood cell count when ANC is greater than or equal to 1500 (alopecia and hypertension exempted).
* Women of childbearing potential must agree to use adequate barrier contraception (interaction with oral contraceptives is unknown) prior to study entry, during therapy and for 3 months after completion of therapy and must have a negative pregnancy test.
* Patients must be able to give written informed consent.

EXCLUSION CRITERIA:

* Evidence of severe or uncontrolled systemic disease or any concurrent condition which in the Investigator's opinion makes it unsafe for the patient to participate in the trial or which would jeopardize compliance with the protocol.
* Evidence of central nervous system (CNS) involvement. Patients with abnormal clinical exam or history will require a head computed tomography (CT) or magnetic resonance imaging (MRI).
* History of clinically symptomatic pancreatitis within the six months prior to enrollment.
* History of prior exposure to any formulation of L-asparaginase.
* Patients with a history of deep venous thrombosis or pulmonary embolism within the past 3 months, or pulmonary embolism within the past 6 months, history of recurrent clot or pulmonary embolism (PE), or those patients requiring ongoing full dose anticoagulation will be ineligible. Line prophylaxis with 1 mg warfarin daily will be allowed.
* Patients with active infection will not be eligible, but may become eligible once infection has resolved and they are at least 7 days from completion of antibiotics.
* Women who are pregnant and women actively breast-feeding will be excluded.
* Previous or current malignancies within the last 5 years, with the exception of cervical carcinoma in situ curatively treated, ductal or lobular carcinoma in situ curatively treated and without ongoing therapeutic intervention, and nonmelanomatous skin cancers curatively treated.
* No concomitant use of complementary or alternative medication or other agents (investigational or anti-cancer agents) will be allowed without approval of a principal investigator (PI) or associate investigator (AI). Every effort will be made to maximize patient safety and minimize changes in chronic medications.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2010-01; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elise C Kohn, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Jemal A, Siegel R, Ward E, Hao Y, Xu J, Murray T, Thun MJ. Cancer statistics, 2008. CA Cancer J Clin. 2008 Mar-Apr;58(2):71-96. doi: 10.3322/CA.2007.0010. Epub 2008 Feb 20. PMID 18287387
- [Background] Liotta LA, Kohn EC. The microenvironment of the tumour-host interface. Nature. 2001 May 17;411(6835):375-9. doi: 10.1038/35077241. PMID 11357145
- [Background] Alvarez AA, Krigman HR, Whitaker RS, Dodge RK, Rodriguez GC. The prognostic significance of angiogenesis in epithelial ovarian carcinoma. Clin Cancer Res. 1999 Mar;5(3):587-91. PMID 10100710
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2010-C-0028.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pegaspargase in Women With Cancer
Started | 4
Completed | 1
Not Completed | 3
Not completed — Death | 1
Not completed — Discontinued study drug | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Pegaspargase in Women With Cancer
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.1 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: 6 Month Progression Free Survival
Description: Proportion of patients able to attain a 6 month progression free survival. Progressive disease is defined as >20% increase in the sum of the longest diameter of all target lesions, or the unequivocal increase in size of non-measurable lesions agreed upon by two investigators, or the appearance of new lesions.
Time Frame: 6 months
Measure: Number; unit: Participants
Arm/Group | Pegaspargase in Women With Cancer
Number analyzed (Participants) | 4
Participants | 0

2. Primary Outcome: Evaluation of Safety in Patients With Ovarian, Fallopian Tube, and/or Primary Peritoneal Cancer.
Description: Here is the number of participants with adverse events. For a detailed list of adverse events see the adverse event module.
Time Frame: 11 months, 25 days
Measure: Number; unit: Participants
Arm/Group | Pegaspargase in Women With Cancer
Number analyzed (Participants) | 4
Participants | 4

ADVERSE EVENTS:
Arm/Group | Pegaspargase in Women With Cancer
Serious Adverse Events (participants affected / at risk) | 2/4
Other Adverse Events (participants affected / at risk) | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pegaspargase in Women With Cancer (N=4)
Allergic reaction (Immune system disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pegaspargase in Women With Cancer (N=4)
Fatigue (General disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (2)
Alkaline phosphatase increased (Investigations) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 2 (2)
Bloating (Gastrointestinal disorders) | 1 (1)
Blood bilirubin increased (Investigations) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fibrinogen decreased (Investigations) | 2 (4)
Gastrointestinal disorders - Other, specify (Urgency bowel movement) (Gastrointestinal disorders) | 1 (1)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (3)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Investigations-Other, specify (PT, high) (Investigations) | 1 (1)
Lipase increased (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Weight loss (Investigations) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No